CLINICAL TRIAL: NCT01390740
Title: Observatory of Screening Aneurysms of the Abdominal Aorta During Echocardiography. National Epidemiological Survey
Acronym: E2T3A
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Serge KOWNATOR, Professor, French Cardiology Society
Other Study IDs: 10 586
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Transthoracic echocardiography
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Echocardiography: patients with echocardiography

SUMMARY:
Study of the prevalence of Abdominal Aortic Aneurysms (AAA) (> 3 cm) in patients with echocardiography (transthoracic or) during a specific day, with cardiologists in France.

This is a cross-sectional epidemiological investigation, assembling evidence from a routine ultrasound screening for AAA at the waning of echocardiograms performed during a specific day.

The study will be offered a list of centers selected by the Scientific Committee in the complete list of locations being in France, the subsidiary of echocardiography Echocardiography of French Society of Cardiology. These centers will be 500 in number representative of the French centers, geographically and by type of centers.

DETAILED DESCRIPTION:
Multicenter observational study collecting data from a routine ultrasound screening for AAA at the waning of echocardiograms performed during a specific day. All of the cardiologists practicing echocardiography are invited to participate in this study, each cardiologist should include echocardiography in 10 patients examined for any reason and will be considered referring cardiologist.

There will be no follow-up, the idea is to have a database with measures of abdominal aortic aneurysms and therefore.

ELIGIBILITY:
Inclusion Criteria:

* Any patient > 65 years,
* Have an echocardiogram, whatever the reason,
* Having agreed to participate in the study.

Exclusion Criteria:

* Patients already operated in the aorta (AAA, PAD, stent, ...)
* Patient refusal to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study proposed a list of centers selected by the Scientific Committee in the complete list of locations being in France, the subsidiary of echocardiography Echocardiography of the French Society of Cardiology. These centers number 500 are representative of the French centers, geographically and by type of centers.
  This is a cross-sectional epidemiological investigation, assembling evidence from a routine ultrasound screening for AAA at the waning of echocardiograms performed during a specific day
Sampling Method: Non-Probability Sample
Enrollment: 1412 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients with AAA among those with echocardiography. | 1 day
  Discovery of the aneurysm of the abdominal aorta at the waning of echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Office of Cardiology Kownator, Thionville, France

REFERENCES:
- [Background] Jaussi A, Fontana P, Mueller XM. Imaging of the abdominal aorta during examination of patients referred for transthoracic echocardiography. Schweiz Med Wochenschr. 1999 Jan 23;129(3):71-6. PMID 10065509
- [Background] Kertai MD, Boersma E, Westerhout CM, van Domburg R, Klein J, Bax JJ, van Urk H, Poldermans D. Association between long-term statin use and mortality after successful abdominal aortic aneurysm surgery. Am J Med. 2004 Jan 15;116(2):96-103. doi: 10.1016/j.amjmed.2003.08.029. PMID 14715323
- [Background] Roshanali F, Mandegar MH, Yousefnia MA, Mohammadi A, Baharvand B. Abdominal aorta screening during transthoracic echocardiography. Echocardiography. 2007 Aug;24(7):685-8. doi: 10.1111/j.1540-8175.2007.00467.x. PMID 17651096
- [Background] Schwartz KV, Rashkow AM, Akella MS. Detection of Abdominal Aortic Aneurysm During Routine Echocardiography. Echocardiography. 1996 Jan;13(1):71-74. doi: 10.1111/j.1540-8175.1996.tb00869.x. PMID 11442905
- [Background] Seelig MH, Malouf YL, Klingler PJ, Oldenburg WA, Atkinson EJ. Clinical utility of routine screening for abdominal aortic aneurysm during echocardiography. Vasa. 2000 Nov;29(4):265-8. doi: 10.1024/0301-1526.29.4.265. PMID 11141649
- [Background] Spittell PC, Ehrsam JE, Anderson L, Seward JB. Screening for abdominal aortic aneurysm during transthoracic echocardiography in a hypertensive patient population. J Am Soc Echocardiogr. 1997 Sep;10(7):722-7. doi: 10.1016/s0894-7317(97)70115-9. PMID 9339423
- [Result] Aboyans V, Bataille V, Bliscaux P, Ederhy S, Filliol D, Honton B, Kurtz B, Messas E, Mohty D, Brochet E, Kownator S; investigators of the E2T3A study. Effectiveness of screening for abdominal aortic aneurysm during echocardiography. Am J Cardiol. 2014 Oct 1;114(7):1100-4. doi: 10.1016/j.amjcard.2014.07.024. Epub 2014 Jul 18. PMID 25127549